CLINICAL TRIAL: NCT05204472
Title: Burst-Deep Brain Stimulation of the Thalamus for Neuropathic Facial Pain and Central Poststroke Pain: a Prospective, Randomized Cross-over Feasibility Trial
Brief Title: Thalamic-Burst-DBS for Neuropathic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DBS for neuropathic pain
Record Dates: First submitted 2022-01-12; First posted 2022-01-24 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Central Post-stroke Pain; Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Burst DBS first, Tonic DBS second (Experimental): 10 days of Burst-stimulation followed by 10 days of active tonic stimulation (Burst-DBS -> tonic-DBS)
  Interventions: Device: Burst DBS; Device: Tonic DBS
- Tonic DBS first, Burst DBS second (Active Comparator): 10 days of active tonic stimulation followed by 10 days of Burst-stimulation (tonic-DBS -> Burst-DBS)
  Interventions: Device: Burst DBS; Device: Tonic DBS

INTERVENTIONS:
Device: Burst DBS — Patients undergo stereotactic implantation of DBS electrodes in the thalamus under local anesthesia. The DBS electrodes will be connected to an external pacemaker for a time period of four weeks. On the first day following surgery, patients will undergo an empirical clinical testing of the stimulation parameter settings. At the same day patients will undergo somatosensory- and contact heat-evoked potential recording for phenotype-stratification (post-hoc analysis).During the next 24 days with the electrodes externalized and connected to the external pacemaker, patients will be randomly assigned in a 1:1 ratio to one of the two groups that undergo two blocks of stimulation:
  12 days of of Burst-stimulation followed by 12 days active tonic stimulation (Burst-DBS -> tonic-DBS) Between each stimulation block the stimulator will be switched off for one day to prevent any hang-over effects of stimulation (wash-out period).
Device: Tonic DBS — Patients undergo stereotactic implantation of DBS electrodes in the thalamus under local anesthesia. The DBS electrodes will be connected to an external pacemaker for a time period of four weeks. On the first day following surgery, patients will undergo an empirical clinical testing of the stimulation parameter settings. At the same day patients will undergo somatosensory- and contact heat-evoked potential recording for phenotype-stratification (post-hoc analysis).During the next 24 days with the electrodes externalized and connected to the external pacemaker, patients will be randomly assigned in a 1:1 ratio to one of the two groups that undergo two blocks of stimulation:
  12 days of active tonic stimulation followed by 12 days of Burst-stimulation (tonic-DBS -> Burst-DBS) Between each stimulation block the stimulator will be switched off for one day to prevent any hang-over effects of stimulation (wash-out period).

SUMMARY:
Central post-stroke pain (CPSP) is a neuropathic pain syndrome and one of the major sequelae after ischemic or hemorrhagic cerebral stroke.

Recently, a modified stimulation paradigm has been developed in the field of spinal cord stimulation (SCS) for a variety of neuropathic pain disorders. To date, this stimulation paradigm has not yet been evaluated systematically for deep brain stimulation to treat neuropathic pain disorders.

The purpose of this clinical investigation is to investigate if Burst-DBS of the thalamus is more effective compared to classical continuous low-frequency stimulation DBS to reduce the subjective pain intensity in patients with chronic neuropathic pain after stroke or in patients with neuropathic facial pain.

DETAILED DESCRIPTION:
Central post-stroke pain (CPSP) is a neuropathic pain syndrome and one of the major sequelae after ischemic or hemorrhagic cerebral stroke. Neuropathic facial pain (NFP) can arise after damage to or affection of the trigeminal nerve caused by trauma, infection or postsurgery and results in characteristic burning and shooting pain of the affected area in the face.

The lack of effective analgesic treatment for these two conditions continues to be an unmet medical need and led to the investigation of alternative treatments of CPSP and NFP such as deep brain stimulation (DBS). DBS is an invasive neuromodulation therapy that consists of placing small electrodes into confined anatomical structures of the brain to deliver small therapeutic currents.

Recently, a modified stimulation paradigm has been developed in the field of spinal cord stimulation (SCS) for a variety of neuropathic pain disorders. This so-called burst stimulation provides pulse trains of five high-frequency pulses at 500 Hz (= 500 Hz spike frequency) occurring 40 times a second (= 40 Hz burst frequency). Burst SCS has been demonstrated to provide a better pain relief compared to classical tonic (continuous application of 50 Hz stimulation) SCS without causing paresthesia. To date, this stimulation paradigm has not yet been evaluated systematically for deep brain stimulation to treat neuropathic pain disorders.

The purpose of this clinical investigation is to investigate if Burst-DBS of the thalamus is more effective compared to classical continuous low-frequency stimulation DBS to reduce the subjective pain intensity in patients with chronic neuropathic pain after stroke or in patients with neuropathic facial pain.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 18-75 years
* Patients suffering from chronic (duration > 12 months) unilateral neuropathic pain caused by an ischemic or haemorrhagic cerebral stroke or
* Patients suffering from chronic (duration > 12 months) unilateral neuropathic facial pain due to one of the following causes:

  1. post-herpes-zoster-neuralgia,
  2. posttraumatic, neuropathic facial pain,
  3. atypical trigeminal neuralgia after surgical intervention
* Severe baseline pain intensity (VAS score > 6/10) considered as resistant to medication specific to neuropathic pain at sufficient doses and durations (including at least antiepileptics and antidepressants)

Exclusion Criteria:

* Significant cognitive impairment (total MOCA score < 1.5 standard deviations from age- and education adapted mean values),
* DSMIV axis I or II psychiatric disorder
* Relevant psychosocial risk factors (any of): history of other chronic pain syndrome, pain catastrophizing, substance abuse, secondary gain
* Contra-indication to surgery, anesthesia, or MRI
* Known or suspected non-compliance or inability to operate the DBS system
* Woman with childbearing potential
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia. etc. of the subject
* Participation in another interventional clinical trial within 30 days prior to this trial or during the trial
* Previous enrollment into the current trial
* Enrolment of the investigator's family members, employees, and other dependent persons
* Patients who are planned to undergo diathermy, electroshock therapy or transcranial magnetic stimulation (TMS)
* Patients with implanted electric devices (i.e. cardiac defibrillator, pacemaker)
* Patients who are at poor surgical risk (i.e. patients with multiple severe illnesses or active general infections)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Percentage reduction of pain intensity | 1 week after surgery
  Percentage reduction of pain intensity on the numeric rating scale (NRS 1-10) after each stimulation-block compared to the baseline pain intensity before surgery. Score 0-10 with 0 representing no pain, and 10 maximum pain intensity
Percentage reduction of pain intensity | 2 weeks after surgery
  Percentage reduction of pain intensity on the numeric rating scale (NRS 1-10) after each stimulation-block compared to the baseline pain intensity before surgery. Score 0-10 with 0 representing no pain, and 10 maximum pain intensity

SECONDARY OUTCOMES:
Change of pain intensity on the numeric rating scale | 12 months after surgery
  Efficacy of DBS after 12 months of open-label stimulation measured as the percentage change of pain intensity on the numeric rating scale compared to baseline. Score 0-10 with 0 representing no pain, and 10 maximum pain intensity
Percentage change of pain intensity on the Neuropathy pain scale | 12 months after surgery
  Efficacy of DBS after 12 months of open-label measured as the percentage change of pain intensity on the Neuropathy pain scale (DN-4) compared to baseline. Score 0-10 with 0 representing no pain, and 100 maximum pain intensity
Percentage improvement of quality of life measured by the EuroQoL 5D-5L | 12 months after surgery
  Efficacy of DBS after 12 months of open-label measured as the percentage improvement of quality of life measured by the EuroQoL 5D-5L questionnaire (Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/ Depression (rating from no problems to extreme problems) and health status self rating by patient (Score 0-100, 0 the worst health and 100 the best health)) compared to baseline.
Change of dosage of analgesic medication(s) | 12 months after surgery
  Change of dosage of analgesic medication(s) at 12 months of open-label stimulation measured as the total dosage in mg per medication per day with reference to baseline
Efficacy of DBS | 12 months after surgery
  Efficacy of DBS after 12 months of open-label stimulation measured as the percentage improvement of depressive symptoms by the BDI questionnaire compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nowacki, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Dep. of Neurosurgery, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No